CLINICAL TRIAL: NCT02245633
Title: Correlation Between Vitamin D Levels to ADAMTS13 , VWF and Micro RNA Expression in Diabetic Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Sydney Ben Shitrit, Dr., Meir Medical Center
Other Study IDs: 0081-14-MMC
Record Dates: First submitted 2014-09-09; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Hemodialysis Patients; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — miRNA will be extract from patient'w plasma

GROUPS / COHORTS (2):
- vitamin D levels deficient: Diabetic hemodialysis patients with vitamin D levels deficient
- vitamin D levels sufficient: Diabetic hemodialysis patients with vitamin D levels sufficient

SUMMARY:
The aim of this research is to study how vitamin D affects various aspects of the disease process, such as inflammation, coagulation (ADAMTS13 and WVF) and miRNAs, in Diabetic kidney disease hemodialysis patients.

Diabetes mellitus (DM) is one of the most common chronic diseases in nearly all countries. Diabetic kidney disease (DKD) traditionally has been referred to as diabetic nephropathy and is one of the microvascular complications of diabetes. Diabetic kidney disease (DKD) occurs in 25%-40% of patients with diabetes .

Some studies have shown that the high risk of cardiovascular disease in diabetic patients with nephropathy is associated with increased plasma levels of von Willebrand factor (VWF) and decreased ADAMTS13 levels. VWF is a glycoprotein that plays an important role in platelet thrombus formation, whereas ADAMTS13 is a proteolytic enzyme that is responsible for degradation of large multimers of VWF released in the plasma by endothelial cells and platelets. Patients with both chronic kidney disease and diabetes have been shown to have higher plasma levels of VWF and decreased ADAMTS13 activity compared to healthy controls.

Increased plasma levels of VWF, which reflects damage to endothelial cells and a hypercoagulability state, have been reported in atherosclerosis and diabetes. Thus, VWF and ADAMTS13 seem to be important players in the interface between diabetic nephropathy, hypercoagulability and atherosclerotic cardiovascular disease. Vitamin D deficiency is a risk factor for DM and hypertension. The investigators previous studies showed that adding calcitriol (activated vitamin D) to endothelial and vascular smooth muscle cells significantly down-regulated the inflammatory response of gene and protein expression involved in the nuclear factor kappa-light-chain-enhancer of activated B cells (NFĸB) signal transduction pathway. Micro RNA (miRNA) are short noncoding RNAs, 22-25 nucleotides long. As an endogenous production transcript, miRNAs can bind to the 3 untranslated regions (3 UTR) of its target messenger RNA (mRNA) in an imperfect, complementary manner, leading to post-transcriptional gene silencing. As a result, miRNAs can inhibit gene expression via mRNA degradation, translation inhibition, or transcriptional inhibition.The critical role of miRNAs has been established in several cellular and biologic processes, such as proliferation, differentiation, and development, and in the regulation of genes related to immune responses, cancer, and insulin secretion. MiRNA are involved in various biological processes and become novel biomarkers, modulators and therapeutic targets for diseases such as cancer, atherosclerosis, and DM.

Significance: The high prevalence of cardiovascular morbidity and mortality in patients with DM on chronic hemodialysis remains a significant clinical problem and the finding of potential new biomarkers should be further investigated. This study aims to establish a link between ADAMTS13, VWF miRNA expression and vitamin D levels that can contribute to the development of new treatments for hemodialysis patients with diabetes.

Methods: Each hemodialysis patient with diabetes in the investigators institute will be asked to participate in the study. After explaining the research goals, patients that agree to participate will sign an informed consent. The investigators estimate that the study will include 70 patients. Each patient will be assessed by a physician and 4 vials of blood will be taken while the patient is connected to the dialysis machine. The blood will be sent to the laboratory to check: 1) chemistry; 2) 1-25 vitamin D and 25- vitamin D levels; 3) ADAMTS13 activity and VWF; and 4) miRNA extraction. The patients will be grouped according to vitamin D levels (deficient /sufficient), and ADAMTS13, VWF and miRNA expression will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic kidney disease - hemodialysis patient with diabetes

Exclusion Criteria:

* Hemodialysis patient - non diabetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients with diabetes at Meir Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-02 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
ADAMTS13 levels in diabetic hemodialysis patients | 1 day
  blood will be collected from diabetic hemodialysis patients that will arrived to the hospital for receive dialysis for analysis ADAMTS13 levels

SECONDARY OUTCOMES:
VWF levels in diabetic hemodialysis patients | 1 day
  blood will be collected from diabetic hemodialysis patients that will arrived to the hospital for receive dialysis for analysis VWF levels

OTHER OUTCOMES:
miRNA expression in plasma from diabetic hemodialysis patients | 1 day
  blood will be collected from diabetic hemodialysis patients that will arrived to the hospital for receive dialysis for extract miRNA

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology dept. Meir Medical Center, Kfar Saba, Israel